CLINICAL TRIAL: NCT05876559
Title: Joyuus: A Web-based Tool for Postpartum Care Self-care to Address the Complex Needs of Underserved Women
Brief Title: Joyuus - A Web-based Tool for Postpartum Care Self-care for Underserved Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joyuus, LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: p-20167; R44MD014923 (NIH)
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Maternal Health
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The investigators plan to conduct a 3-month, parallel-group, randomized controlled trial (RCT) to evaluate the effectiveness on improving maternal functioning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active intervention group (Experimental): Participants will receive immediate access to Joyuus selfcare mobile app
  Interventions: Other: Joyuus Self-care Mobile App
- standard care control group (Active Comparator): Participants will receive standard care, and will not have access to Joyuus selfcare mobile app until study completion.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Joyuus Self-care Mobile App — Joyuus is an innovative self-care mobile tool designed to address the needs of underserved women who are at greater risk for adverse postpartum outcomes. It provides the appropriate information, knowledge, and skills to improve postpartum health through self-care, and identifies when it is appropriate to seek care.
  Arms: active intervention group
Other: Standard Care — Standard care is access to typical resources women have access to during postpartum and does not include the Joyuus intervention.
  Arms: standard care control group

SUMMARY:
The goal of this RCT is to evaluate the effectiveness of Joyuus on improving maternal functioning with postpartum moms. The main questions it aims to answer are:

* The primary hypothesis is that participants of the Joyuus program will demonstrate improved functional status compared to the control arm participants at 3-month follow-up.
* The secondary hypotheses are that participants using the Joyuus tool will demonstrate improvement in depression, anxiety, resilience, social support, and knowledge compared to the control arm at 6- and 12-weeks follow-up.

DETAILED DESCRIPTION:
In the United States, the postpartum period is a critical time for both maternal and child health; the US maternal mortality rate is the highest among other developed, high-income countries. More than half of all maternal deaths occur postpartum, from one day to one year after birth. There are vast racial and ethnic disparities in maternal mortality and severe morbidity, disproportionately experienced by Black and Latina mothers and other BIPOC women. Black women are 3-4 times more likely to experience maternal mortality than white women10, and Hispanic women are twice as likely to experience severe maternal outcomes compared with non-Hispanic white women. The American College of Obstetricians and Gynecologists recognized the deficiencies in postpartum care and coined the term the 'fourth trimester' to mark the time following birth through the first 3-months postpartum. They recently updated recommendations to address these challenges. The Biden Build Back Better Act also prioritized this issue. Joyuus is a web-based self-care mobile tool addressing the 12 months postpartum, to reduce the risks of avoidable morbidity and mortality for underserved women. The tool addresses physical, mental, real world, cultural, and knowledge barriers which impact quality postpartum care. Joyuus provides information, resources, expert perspectives, peer communications and red flags presented in a variety of formats to help women identify how to adopt healthy self-care habits. Importantly, it also identifies when self-care leads to seeking provider care. Pregnant women often turn to the internet to find information about their health and their developing baby's health. Yet, studies find that mothers are not finding sufficient resources to match their postpartum needs. The Phase I grant demonstrated in a sample of Black women that this audience is highly engaged across the income and education spectrum and prefers mobile access and text-based communication. In Phase II work will continue to include lived experiences of women most at risk for negative postpartum outcomes as part of the complete tool. The first step will be to conduct a needs assessment to understand informational, cultural and language wants and needs in the Latina population. The broader randomized trial will invite a diverse population of BIPOC and white women. The Phase II scope aims to complete three major tasks:

AIM 1: Expand feasibility activities to address Latina population. Explore self-care (and seeking care) needs for the postpartum Latina community and integrate with the Phase I focus group findings.

AIM 2: Build complete tool. The investigators will complete the development of a fully interactive Joyuus web based mobile tool in English and Spanish.

AIM 3: Test in randomized controlled trial. The investigators will test the effectiveness of Joyuus with a diverse national sample of postpartum women, considering the impact on maternal function, depression, anxiety, resilience, knowledge, and social support.

ELIGIBILITY:
Inclusion Criteria:

* Must be age 18 or older
* Must be between 0-6 months postpartum
* Must have a smartphone with internet access and are willing to use this device to participate in all study activities; and
* Must be able to speak, read, and write in English

Exclusion Criteria:

* Medical/health issues which would impact participants' health or ability to participate
* Did not have a live birth

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is about postpartum health for mothers who have given birth. The study does not distinguish on gender identity but focuses on birthing people.
Enrollment: 137 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Barkin Index of Maternal Functioning (BIMF) | Change between baseline and 12 months
  The BIMF is a 20-item self-report measure designed to assess overall functioning in the context of new motherhood. Functional domains include social support, management, mother-child interaction, infant care, self-care, adjustment, and psychological well-being (of the mother). The BIMF demonstrates strong internal consistency. with Cronbach's alpha for the full 20-item scale between .83-.87 indicating strong inter-item agreement. A total score is generated from summing the 20 items (after the reverse-coding of items 16 and 18) and ranges from 0 to 120. Higher total scores are associated with greater levels of functioning.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | Change between baseline and 12 months
  (EPDS), a reliable, valid, and widely used scale that measures the presence and intensity of depressive symptoms. The scale has high internal consistency, test-retest reliability, and construct validity. Each answer is given a score of 0 to 3. The total scores are calculated with a maximum score of 30. Lower scores indicate lower presence or intensity.
State-Trait Anxiety Inventory (STAI) | Change between baseline and 12 months
  The STAI has 20 items for assessing trait anxiety and 20 for state anxiety. Considerable evidence attests to the reliability and validity of the scale. Each type of anxiety has its own scale of 20 different questions that are scored. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Connor-Davidson Resilience Scale (CDRS) | Change between baseline and 12 months
  The CDRS is a 25-item scale covering 17 resilience domains and used across languages, racial/ethnic, and cultural groups. It has been shown to have strong psychometric properties and has validated short forms. CDRS uses a scale of 0-4 with 0 being not true at all, to 4 being true nearly all the time.

OTHER OUTCOMES:
COVID-19 and Mental Health Impacts Scale | Change between baseline and 12 months
  While not a formal endpoint, a descriptive analysis of this measure will be conducted. The COVID-19 Community Response Survey, Mental Health Impact Module is a 13-item questionnaire that was developed to better understand people's experiences about how their lives have changed as a result of COVID-19. Question 1 is a four point scale from Not at all, to 5-7 days. More days indicates increased impact. Questions 2-13 are scored on a 5 point scale from Strongly Disagree to Strongly Agree, with stronger agreement indicating increased impact.
Maternal Health Knowledge | Change between baseline and 12 months
  Knowledge will be assessed by a brief study-specific multiple-choice instrument, to be developed as part of this modest trial, and designed to test understanding of evidence-based concepts presented in the Joyuus tool. While not a formal endpoint, a descriptive analysis of this measure will be conducted. Questions will be scored on a 5 point scale from Strongly Disagree to Strongly Agree, with stronger agreement indicating increased knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Lisa Marceau, Westerly, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No